CLINICAL TRIAL: NCT02715908
Title: A Extension Clinical Study to Evaluate the Long-term Safety and Efficacy of LBEC0101 When Co-administered With Methotrexate (MTX) for Additional 48 Weeks in Patients With RA Who Have Completed the Treatment Period of LG-ECCL002
Brief Title: A Study to Evaluate the Long-term Safety and Efficacy of LBEC0101 in Subjects With Active RA Despite Methotrexate (MTX)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-ECCL004
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — LBEC0101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LBEC0101 (Experimental): Etanercept 50mg
  Interventions: Drug: LBEC0101

INTERVENTIONS:
Drug: LBEC0101 — Etanercept 50mg

SUMMARY:
To evaluate the long-term safety including immunogenicity and efficacy of LBEC0101 50 mg subcutaneous weekly injection when co-administered with MTX

DETAILED DESCRIPTION:
this study is to evaluate the long-term safety including immunogenicity and efficacy of LBEC0101 50 mg subcutaneous weekly injection when co-administered with MTX for additional 48 weeks (a total of 100 weeks including 52 weeks of the treatment period in Study LG-ECCL002) in the subjects who have completed the treatment period of phase III clinical study for LBEC0101 (Study No. LG-ECCL002).

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the treatment period of Study LG-ECCL002
* Patients requiring continuous treatment for rheumatoid arthritis upon the investigator's discretion
* For childbearing female patients or surgically non-sterile male patients, those who agreed to avoid pregnancy using proper contraceptive methods during the study.
* Patients who made a voluntary decision to participate in this clinical study and gave a voluntary written consent to comply with all the instructions with full understanding after being informed of the study

Exclusion Criteria:

* Patients deemed difficult to participate in this extension study due to the adverse events which occurred in Study LG-ECCL002, upon the investigator's discretion at screening
* Patients with at least 10 swollen joints (out of the total 66 assessing joints) or at least 12 tender joints (out of the total 68 assessing joints) at screening
* Women in pregnancy or lactation, or patients planning to be pregnant during the study period
* Patients ineligible for this clinical study upon the investigator's discretion

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
DAS28-ESR | 48 weeks
  Mean change in DAS28-ESR score from baseline (Weeks 0 and 52) at Weeks 76 and 100

SECONDARY OUTCOMES:
DAS28-CRP | 48 weeks
  Mean change in DAS28-CRP score from baseline (Weeks 0 and 52) at Weeks 76 and 100
ACR 20, 50, 70 | 48 weeks
  Response rate on ACR20, 50, 70 at Weeks 52, 76, and 100 based on baseline (Week 0)
Remission rate | 48 weeks
  Remission rate (i.e., DAS28-ESR <2.6) at Weeks 52, 76, and 100
EULAR response | 48 weeks
  Rate of EULAR response on DAS28-ESR at Weeks 52, 76, and 100

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park MC, Matsuno H, Kim J, Park SH, Lee SH, Park YB, Lee YJ, Lee SI, Park W, Sheen DH, Choe JY, Choi CB, Hong SJ, Suh CH, Lee SS, Cha HS, Yoo B, Hur JW, Kim GT, Yoo WH, Baek HJ, Shin K, Shim SC, Yang HI, Kim HA, Park KS, Choi IA, Lee J, Tomomitsu M, Shin S, Lee J, Song YW. Long-term efficacy, safety and immunogenicity in patients with rheumatoid arthritis continuing on an etanercept biosimilar (LBEC0101) or switching from reference etanercept to LBEC0101: an open-label extension of a phase III multicentre, randomised, double-blind, parallel-group study. Arthritis Res Ther. 2019 May 21;21(1):122. doi: 10.1186/s13075-019-1910-2. PMID 31113455